CLINICAL TRIAL: NCT05813626
Title: Neoadjuvant Chemotherapy Plus Toripalimab in Patients With Locoregionally Advanced Nasopharyngeal Carcinoma
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Zhejiang Cancer Hospital (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: NPC-202301
Record Dates: First submitted 2023-03-06; First posted 2023-04-14 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-03

CONDITIONS: Nasopharyngeal Carcinoma
MeSH Terms: conditions — Nasopharyngeal Carcinoma | interventions — toripalimab

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- Toripalimab Combined with Induction Chemotherapy (Experimental): Induction chemotherapy (IC; every 3 weeks × 3 cycles; gemcitabine 1000 mg/m2 day 1, 8 + cisplatin 80 mg/m2 day 1); Toripalimab, 240 mg, day 1; start on day 1 of the first cycle IC and continue every 3 weeks for 3 cycles till the end of IC.
  Interventions: Drug: Toripalimab

INTERVENTIONS:
Drug: Toripalimab — Toripalimab (240 mg Q3W for 3 cycles) combine with chemotherapy

SUMMARY:
Neoadjuvant chemotherapy plus toripalimab in patients with locoregionally advanced nasopharyngeal carcinoma

ELIGIBILITY:
Inclusion Criteria:

1. Age: 18 to 65;
2. Pathological type: non-keratinizing carcinoma (World Health Organization criteria);
3. Diagnosed with LANPC according to the 8th edition clinical staging system of the American Joint Committee on Cancer [AJCC]/Union for International Cancer Control [UICC];
4. ECOG performance score: 0 to 1;
5. Normal bone marrow function: white blood cell count > 4×109/L, hemoglobin > 90g/L, platelet count > 100×109/L;
6. Normal values of thyroid function, amylase and lipase examination, pituitary function, inflammation and infection indicators, myocardial enzymes, and ECG results. For patients older than 50 years with a smoking history, normal lung function are required. Patients with abnormal ECG and/or a history of vascular disease (but not meeting the exclusion criteria listed in the exclusion criteria 7) need further testing and require normal results of myocardial function and color Doppler ultrasound.
7. Normal liver and kidney function: total bilirubin ≤ 1.5 × upper limit of normal (ULN); alanine transaminase and aspartate transaminase ≤ 2.5 × ULN; alkaline phosphatase ≤ 2.5 × ULN; creatinine clearance rate ≥ 60 ml/min;
8. Patients must sign informed consent and be willing and able to comply with the requirements of visits, treatment, laboratory tests and other research requirements stipulated in the research schedule;
9. Subjects with pregnancy ability must agree to use reliable contraceptive measures from screening to 1 year after treatment.

Exclusion Criteria:

1. Hepatitis B virus surface antigen (HBsAg) positive and HBV DNA > 1×10E3 copies/ml; anti-hepatitis C virus positive;
2. Anti-human immunodeficiency virus (HIV) positive or diagnosed with acquired immune deficiency syndrome (AIDS);
3. Active tuberculosis: active tuberculosis in the past 1 year should be excluded regardless with treatment; history of active tuberculosis over 1 year should be excluded except that previous regulatory anti-tuberculosis treatment is proved;
4. Active, known or suspected autoimmune disease (including but not limited to uveitis, enteritis, hepatitis, pituitary, nephritis, vasculitis, hyperthyroidism, hypothyroidism and asthma requiring bronchiectasis). Exceptions are type I diabetes mellitus, hypothyroidism requiring hormone replacement therapy, skin disorders requiring no systemic treatment (such as vitiligo, psoriasis or alopecia);
5. Previous interstitial lung disease or pneumonia requiring oral or intravenous steroid therapy;
6. Chronic treatment with systemic glucocorticoid (dose equivalent to or over 10 mg prednisone per day) or any other form of immunosuppressive therapy. Subjects who used inhaled or topical corticosteroids were eligible;
7. Uncontrolled heart disease, for example: 1) heart failure (NYHA level ≥ 2); 2) unstable angina; 3) myocardial infarction in past 1 year; 4) supraventricular or ventricular arrhythmia requiring treatment or intervention;
8. Pregnant or lactating women (pregnancy test should be considered for women with sexual life and fertility);
9. Previous or concurrent with other malignant tumors, except for adequately treated non-melanoma skin cancer, cervical carcinoma in situ and thyroid papillary cancer;
10. Allergy to macromolecular protein preparations, or any component of nivolumab;
11. Active infection requiring systemic treatment;
12. Receiving live vaccine within 30 days of the initial nivolumab;
13. History of organ transplantation;
14. History of psychotropic disease, alcoholism or drug abuse; other situation assessed by the investigators that may compromise the safety or compliance of patients, such as serious disease requiring timely treatment (including mental illness), severe laboratory abnormalities, or family-social risk factors.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 89 (Estimated)
Dates: Start 2023-04-03 (Estimated); Primary Completion 2024-10-30 (Estimated); Study Completion 2027-10-30 (Estimated)

PRIMARY OUTCOMES:
Complete Response | 9 weeks
  CR assessed by investigator, according to the Response Evaluation Criteria in Solid Tumors (RECIST1.1) from the National Cancer Institute (NCI). Complete response defined as the complete disappearance of the target and non-target lesion(s) identified at baseline after radiological evaluation by Magnetic Resonance Imaging.

SECONDARY OUTCOMES:
Overall Survival(OS) | 3 years
  defined as the time from random assignment to death from any cause or censored at the date of last follow-up.
Locoregional failure-free survival(LRRFS) | 3 years
  defined as the time from random assignment to local or regional relapse, or death from any cause.
Distant metastasis-free survival(DMFS) | 3 years
  defined as the time from random assignment to distant metastasis, or death from any cause.
Number of participants with adverse events | up to 3 years
  Numbers of patients of treatment-related adverse events were assessed by CTCAE v5.0.
Quality of life (QoL): questionnaire | Week 1,9,16,28
  QoL is evaluated with the use of the head-and-neck-specific module (H&N35) of the Quality of Life Questionnaire-Core 30 module (QLQ-C30), which is established by European Organization for Research and Treatment of Cancer (EORTC). Scores for the module range of H&N35 QLQ-C30 from 0 to 100, with higher scores indicating better functioning or well-being or higher symptom burden (scales measuring symptom burden were reverse-scored to facilitate presentation)

CONTACTS AND LOCATIONS:
Locations (1):
- Zhejiang Cancer Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: Yes